CLINICAL TRIAL: NCT00382473
Title: Mitochondrial Dysfunction in Type 2 Diabetes Mellitus and Capacity for Fat Oxidation During Exercise
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of funding
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 0605115
Record Dates: First submitted 2006-09-28; First posted 2006-09-29 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-04

CONDITIONS: Diabetes Mellitus, Type 2; Overweight
Keywords: Diabetes Mellitus, Type 2; Overweight; Fatty acid oxidation; Mitochondria; Exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- exercise (Experimental)
  Interventions: Behavioral: Aerobic exercise program - 8 weeks

INTERVENTIONS:
Behavioral: Aerobic exercise program - 8 weeks — No drugs. Regular aerobic exercise in structured prescription format

SUMMARY:
The purpose of this study is to compare the effects of an 8-week aerobic training program upon fat oxidation in vivo and markers of skeletal muscle mitochondrial content and oxidative capacity in sedentary obese subjects with and without type 2 diabetes. We will also investigate if mitochondrial content in muscle predicts success of weight loss.

The specific aims are:

* To compare systemic fat oxidation rates;
* To measure mitochondrial content in muscle before and after aerobic training;
* To determine if decreased mitochondrial content is also associated with decreased mitochondrial oxidative capacity;
* To measure non-plasma fatty acid oxidation in vivo during submaximal exercise conditions both prior and after aerobic training;
* To determine whether increases in fat oxidation due to physical activity predict weight loss success when a reduced calorie diet is added to a physical activity program.

DETAILED DESCRIPTION:
During prolonged moderate-intensity exercise, skeletal muscle gradually increases its metabolic reliance on fat oxidation. In healthy subjects, this adaptation is enhanced by aerobic training and is associated with increased mitochondrial capacity in muscle. Whether or not subjects with type-2 diabetes (T2DM) respond to exercise training with similar metabolic and mitochondrial adaptations is yet to be demonstrated. Skeletal muscle mitochondrial oxidative capacity has been shown to be deficient in T2DM, suggesting a compromised physiologic reserve that might have implications for the metabolic plasticity of muscle during exercise.

This study will test the hypothesis that fat oxidation rates during exercise are poorly responsive to training in T2DM, being correlated to the degree of muscle mitochondrial adaptation. The effects of a 16-week intervention (8 weeks of exercise intervention followed by 10-12 weeks of weight loss intervention) on systemic fat oxidation during exercise and mitochondrial capacity will be compared between 3 sedentary subject groups; 15 lean subjects, 15 overweight subjects with T2DM, and 15 overweight subjects without diabetes. The first aim is to compare the degree of improvement in fat oxidation during submaximal exercise obtained by indirect calorimetry. The second and third aims are, respectively, to compare the degree of improvement in mitochondrial content and oxidative capacity in muscle biopsy samples. The fourth aim is to determine whether fat oxidation from non-plasma sources is increased by the intervention. The final aim is to examine whether improvements in fat oxidation predict degree off success in a subsequent weight loss program.

The results of this study will be relevant to the understanding of the mechanisms by which exercise training confers metabolic improvements in T2DM. In addition, this study will address whether perturbations in mitochondria could explain why obese individuals with T2DM might have difficulty with fat disposal.

ELIGIBILITY:
Inclusion Criteria:

Men and women, aged 28-55 year-old, in general good health and with no contraindications to exercise. We are recruiting three groups of subjects: Group 1: overweight/obese adults with type 2 diabetes, with a BMI between 28-40. Group 2: overweight/obese adults without type 2 diabetes, with a BMI between 28-40. Group 3: adults without type 2 diabetes, with a BMI equal or less than 25 (not overweight/obese.)

Exclusion Criteria:

Any condition that does not permit exercise; current participation in a regular physical activity; uncontrolled blood pressure; treatment with any of the following medications: insulin, any weight-loss drug, oral glucocorticoids, or any drugs that affect muscle and fat metabolism such as niacin, fibrates, and beta blockers

Ages: 28 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2006-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The degree of improvement in fat oxidation during submaximal exercise obtained by indirect calorimetry after subjects have completed an eight week aerobic exercise program. | 8 weeks

SECONDARY OUTCOMES:
The degree of improvement in muscle mitochondrial content after eight week exercise program. | 8 weeks
The amount of improvement in muscle mitochondrial oxidative capacity after eight week exercise program. | 8 weeks
Increase in fat oxidation from non-plasma sources after the eight week intervention. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Frederico G Toledo, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Montefiore Hospital, Pittsburgh, Pennsylvania, United States